CLINICAL TRIAL: NCT06004050
Title: A Phase 3 Trial to Evaluate Efficacy, Safety, and Pharmacokinetics of Twice-Daily Applications of Delgocitinib Cream 20 mg/g in Chinese Adults and Adolescents (12-17 Years of Age) With Moderate to Severe Chronic Hand Eczema
Brief Title: A Trial to Evaluate Efficacy, Safety, and Pharmacokinetics of Delgocitinib Cream in Chinese Adults and Adolescents With Moderate to Severe Chronic Hand Eczema
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LP0133-2283
Record Dates: First submitted 2023-08-16; First posted 2023-08-22 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-07

CONDITIONS: Chronic Hand Eczema
Keywords: Dermatologic Disease; Dermatology; Eczema; Chronic Hand Eczema; Delgocitinib
MeSH Terms: conditions — Skin Diseases; Eczema | interventions — delgocitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Double-Blind Period: Twice-Daily Delgocitinib Cream (Experimental): 20 mg/g twice daily
  Interventions: Drug: Delgocitinib
- Double-Blind Period: Twice-Daily Vehicle Cream (Placebo Comparator): 20 mg/g twice daily
  Interventions: Other: Vehicle cream
- Open Label Period: Twice-Daily Delgocitinib (Experimental): 20 mg/g twice daily
  Interventions: Drug: Delgocitinib

INTERVENTIONS:
Drug: Delgocitinib — Topical administration
  Arms: Double-Blind Period: Twice-Daily Delgocitinib Cream; Open Label Period: Twice-Daily Delgocitinib
Other: Vehicle cream — Topical administration
  Arms: Double-Blind Period: Twice-Daily Vehicle Cream

SUMMARY:
The primary objective of this study is to evaluate the efficacy of twice-daily applications of delgocitinib cream 20 mg/g compared with cream vehicle in the treatment of participants with moderate to severe chronic hand eczema (CHE).

DETAILED DESCRIPTION:
The trial comprises of a 16-week double-blind, treatment period, followed by an open label treatment period of 36 weeks. In the double-blind treatment period two thirds of participants will be randomly assigned to receive delgocitinib and one third will receive placebo/vehicle. In the double-blind treatment period, participants will use delgocitinib twice a day. In the open label period, participants will only use delgocitinib when needed (if their CHE flares up). Some participants will also give blood samples at the start of the trial for pharmacokinetic measurements. Participants will visit the clinic every 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or above at screening for adult participants and age 12-17 years at screening and baseline for adolescent participants.
2. Diagnosis of CHE, defined as hand eczema that has persisted for more than 3 months or returned twice or more within the last 12 months. Disease severity graded as moderate to severe at screening and baseline according to IGA-CHE (i.e. an IGA-CHE score of 3 or 4).
3. HESD itch score (weekly average) of ≥4 points at baseline. The baseline weekly average will be calculated from daily assessments of itch severity during the 7 days immediately preceding the baseline visit (Day -7 to Day -1). A minimum of 4 itch scores out of the 7 days is required to calculate the baseline average score.
4. Participants who have a documented recent history of inadequate response to treatment with topical corticosteroids (TCS) (at any time within 1 year before the screening visit) or for whom TCS are documented to be otherwise medically inadvisable (e.g. due to important side effects or safety risks).

   * Inadequate response is defined as a history of failure to achieve and maintain a low disease activity state (comparable to an IGACHE score of ≤2) despite treatment with a daily regimen of TCS of class III-IV (potent to very potent), applied for at least 28 days or for the maximum duration recommended by the product prescribing information, whichever is shorter.
   * Important side effects or safety risks are those that outweigh the potential treatment benefits and include intolerance to treatment, hypersensitivity reactions, and significant skin atrophy as assessed by the physician.
5. Participants adherent to standard non-medicated skin care including avoidance of known and relevant irritants and allergens.
6. A woman of childbearing potential (WOCBP) must use an acceptable method of birth control throughout the trial up until the last application of investigational medicinal product (IMP).

Exclusion Criteria:

1. Active atopic dermatitis (AD) requiring medical treatment in regions other than the hands and feet.
2. Hyperkeratotic hand eczema in combination with a history of psoriasis on any part of the body.
3. Clinically significant infection (e.g. impetiginized hand eczema) on the hands.
4. Clinically significant infection within 28 days prior to baseline which, in the opinion of the investigator, may compromise the safety of the participant in the trial, interfere with evaluation of the investigational medicinal product (IMP), or reduce the participant's ability to participate in the trial. Clinically significant infections are defined as:

   * A systemic infection.
   * A serious skin infection requiring parenteral (intravenous or intramuscular) antibiotics, antiviral, or antifungal medication.
5. History of any known primary immunodeficiency disorder including a positive human immunodeficiency virus (HIV) test at screening, or the participant taking antiretroviral medications as determined by medical history and/or participant's verbal report.
6. History of cancer:

   * Participants who have had basal cell carcinoma, localized squamous cell carcinoma of the skin or in situ carcinoma of the cervix are eligible provided that the participant is in remission and curative therapy was completed at least 12 months prior to screening.
   * Participants who have had other malignancies are eligible provided that the participant is in remission and curative therapy was completed at least 5 years prior to screening.
7. Any disorder which is not stable and could:

   * Affect the safety of the participant throughout the trial.
   * Impede the participant's ability to complete the trial. Examples include but are not limited to cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, hematologic, immunological, and psychiatric disorders, and major physical impairment.
8. Any abnormal finding which may:

   * Put the participant at risk because of their participation in the trial.
   * Influence the participant's ability to complete the trial. The abnormal finding must be clinically significant and observed during the screening period. Examples include abnormal findings in physical examination, vital signs, ECG, hematology, clinical chemistry, or urinalysis.
9. Positive hepatitis B surface antigen or hepatitis C virus antibody serology at screening.
10. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) level ≥2.0×ULN at screening.
11. Known or suspected hypersensitivity to any component(s) of the IMP.
12. Systemic treatment with immunosuppressive drugs (e.g. methotrexate, cyclosporine, azathioprine), immunomodulating drugs, retinoids (e.g. alitretinoin), traditional Chinese medicines (TCMs) (including herbals), or corticosteroids within 28 days prior to baseline (steroid eyedrops and inhaled or intranasal steroids corresponding to up to 1 mg prednisolone for allergic conjunctivitis, asthma, or rhinitis are allowed).
13. Use of tanning beds, phototherapy (e.g. UVB, UVA1, PUVA), or bleach baths on the handswithin 28 days prior to baseline.
14. Previous or current treatment with Janus Kinase (JAK) inhibitors (including delgocitinib/LEO 124249),systemic or topical.
15. Cutaneously applied treatment with immunomodulators (e.g. PDE-4 inhibitors, pimecrolimus, tacrolimus), TCMs (including herbals), or TCS on the hands within 14 days prior to baseline.
16. Use of systemic antibiotics or cutaneously applied antibiotics on the hands within 14 days prior to baseline.
17. Other transdermal or cutaneously applied therapy on the hands (except for the use of participant's own emollients) within 7 days prior to baseline.
18. Cutaneously applied treatments in regions other than the hands, which could interfere with clinical trial evaluations or pose a safety concern within 7 days prior to baseline.
19. Treatment with any marketed biological therapy or investigational biologic agents (including immunoglobulin, anti-IgE, and dupilumab):

    • Any cell-depleting agents including but not limited to rituximab: within 6 months prior to baseline, or until lymphocyte count returns to normal, whichever is longer.

    • Other biologics: within 3 months or 5 half-lives, whichever is longer, prior to baseline.
20. Treatment with any non-marketed drug substance (that is, an agent that has not yet been made available for clinical use following registration) within the last 28 days prior to baseline or 5 half-lives, whichever is longer.
21. Major surgery within 8 weeks prior to screening, or planned in-patient surgery or hospitalization during the trial period.
22. Current participation in any other interventional clinical trial.
23. Previously randomized in this clinical trial.
24. Concurrent skin diseases on the hands, e.g. tinea manuum.
25. Active psoriasis on any part of the body.
26. Current or recent chronic alcohol or drug abuse, or any other condition associated with poor compliance as judged by the investigator.
27. Employees of the trial site, or any other individuals directly involved with the planning or conduct of the trial, or immediate family members of such individuals.
28. Participants who are legally institutionalized.
29. Women who are pregnant or lactating.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 362 (Actual)
Dates: Start 2023-09-05 (Actual); Primary Completion 2024-12-16 (Actual); Study Completion 2025-09-12 (Actual)

PRIMARY OUTCOMES:
Investigator Global Assessment for Chronic Hand Eczema Score (IGA-CHE TS) at Week 16 | Week 16
  The IGA-CHE score ranges from 0 (clear) to 4 (severe). Treatment response is defined as a score of 0 or 1.

SECONDARY OUTCOMES:
Hand Eczema Severity Index (HECSI)-90 at Week 16 | Week 16
  Defined as at least a 90% improvement in HECSI score from baseline.
HECSI-75 at Week 16 | Week 16
  Defined as at least a 75% improvement in HECSI score from baseline.
Percentage Change in HECSI Score From Baseline to Week 16 | Baseline and Week 16
  HECSI score is used to rate the severity of hand eczema and ranges from 0 (lowest possible score) to 360 (highest possible score).
Number of Participants With Reduction of Hand Eczema Symptom Diary (HESD) Itch Score by ≥4 Points From Baseline at Week 16 | Baseline and Week 16
Number of Participants With Reduction of HESD Score by ≥4 Points From Baseline at Week 16 | Baseline and Week 16
Number of Participants With Reduction of HESD Pain Score by ≥4 Points From Baseline at Week 16 | Baseline and Week 16
Change in Dermatology Life Quality Index (DLQI) Score From Baseline to Week 16 | Baseline and Week 16
Change in HESD Score From Baseline to Week 16 | Baseline and Week 16
Change in HESD Itch Score From Baseline to Week 16 | Baseline and Week 16
Change in HESD Pain Score From Baseline to Week 16 | Baseline and Week 16
Change in Hand Eczema Impact Scale (HEIS) Score | Baseline and Week 16
Change in HEIS Proximal Daily Activity Limitations (PDAL) Score | Baseline and Week 16
Number of Participants With Reduction of DLQI Score of ≥4 Points From Baseline at Week 16 | Baseline and Week 16
Number of Treatment-Emergent Adverse Events (AEs) | From baseline to Week 16
Number of Treatment-Emergent AEs | From Week 16 to Week 54
Area Under the Curve (AUC 0-12) | Day 1 and Day 8 post-dose
Maximum Serum Concentration (Cmax) | Day 1 and Day 8 (0-12 hours post-dose)
Time to Peak Drug Concentration (Tmax) | Day 1 and Day 8 (0-12 hours post-dose)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — LEO Pharma
Locations (24):
- China (24):
  - LEO Pharma Investigational Site, Beijing
  - LEO Pharma Investigational Site, Changchun
  - LEO Pharma Investigational Site, Changsha
  - LEO Pharma Investigational Site, Changzhou
  - LEO Pharma Investigational Site, Chengdu
  - LEO Pharma Investigational Site, Fuzhou
  - LEO Pharma Investigational Site, Guangzhou
  - LEO Pharma Investigational Site, Guiyang
  - LEO Pharma Investigational Site, Hangzhou
  - LEO Pharma Investigational Site, Hefei
  - LEO Pharma Investigational Site, Nanchang
  - LEO Pharma Investigational Site, Nanjing
  - LEO Pharma Investigational Site, Nanyang
  - LEO Pharma Investigational Site, Shanghai
  - LEO Pharma Investigational Site, Shenyang
  - LEO Pharma Investigational Site, Shenzhen
  - LEO Pharma Investigational Site, Shijiazhuang
  - LEO Pharma Investigational Site, Wenzhou
  - LEO Pharma Investigational Site, Wuhan
  - LEO Pharma Investigational Site, Wuxi
  - LEO Pharma Investigational Site, Xianyang
  - LEO Pharma Investigational Site, Yinchuan
  - LEO Pharma Investigational Site, Yiwu
  - LEO Pharma Investigational Site, Zhenjiang

IPD SHARING:
Plan to Share IPD: No